CLINICAL TRIAL: NCT05791448
Title: First in Human Dose Escalation Study of AU409 in Patients With Advanced Primary Liver Cancers or Advanced Solid Tumor With Liver Predominant Metastatic Disease
Brief Title: AU409 for the Treatment of Advanced Primary Liver Cancers or Solid Tumor With Liver Metastatic Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Auransa, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-22-19; NCI-2023-01399 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0C-22-19 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cholangiocarcinoma; Advanced Hepatocellular Carcinoma; Advanced Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Liver; Refractory Malignant Solid Neoplasm; Stage III Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (AU409) (Experimental): Patients receive AU409 PO on study. Patients also undergo CT or MRI and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: RNA Transcription Modulator AU-409

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: RNA Transcription Modulator AU-409 — Given PO
  Other Names: AU 409; AU-409; AU409

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of a new intervention, AU409, in treating patients with primary liver cancers that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or advanced solid tumors that have spread to the liver (liver metastatic disease). AU409 may stop cancer from growing and spreading. This trial may help researchers determine if AU409 is safe and effective in treating patients with liver cancers and solid tumors with liver metastatic disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine maximum tolerated dose (MTD) of RNA transcription modulator AU-409 (AU409) and the recommended phase II dose (RP2D).

II. To characterize the safety and tolerability of AU409 by assessing toxicities per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 criteria.

SECONDARY OBJECTIVES:

I. To obtain a preliminary assessment of anti-tumor activity of AU409 via objective radiologic response using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

II. To determine pharmacokinetics of AU409 in patients with advanced-stage solid tumors.

EXPLORATORY OBJECTIVES:

I. To evaluate the concentration of AU409 in tumor tissue from liver biopsy samples obtained from a subset of patients treated with AU409 at dose level 4 (300 mg) and above.

II. To evaluate expression of genes with TATA box promotion regions on pre- and post- treatment liver biopsy samples.

OUTLINE: This is a dose-escalation study.

Patients receive AU409 orally (PO) on study. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and collection of blood samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Patients must have histopathologically /cytologically confirmed advanced solid tumor, which is refractory to standard therapeutic options, or for which there are no standard therapeutic options. Failure of all approved therapies that have a marginal impact on survival is not required as long as the treating physician considers that treatment on study is appropriate for the subject and documents that the subject elects to defer the approved therapies
* During the dose-escalation portion, patients must have primary liver malignancy (including hepatocellular carcinoma or cholangiocarcinoma) OR a solid tumor with liver dominant disease; liver dominant disease is defined as the majority of the tumor burden being in the liver per investigator assessment AND no more than two extrahepatic sites of disease (site of disease refers to organ or system). During the dose expansion portion of the study, eligibility may be limited to one or more tumor types depending on findings from the dose-escalation phase; this will be clarified in an amendment
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient must have recovered from any toxic effects of previous chemotherapy, targeted therapy or radiotherapy as judged by the Investigator to =< grade 1 (except for alopecia). Residual sensory neuropathy =< grade 2 is allowed. Residual endocrine adverse events (such as hypothyroidism or hypoadrenalism) that are manageable with replacement therapy are allowed
* Previous chemotherapy/radiotherapy/targeted/immunotherapy therapy should have been completed at least 4 weeks prior to start of AU409 administration, or five half-lives, whichever is shorter (except for palliative radiation therapy that should be completed >= 14 days prior to study entry)
* Patients must have an estimated life expectancy of at least 3 months
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation. A male participant must agree to use highly effective contraception during the intervention period and for 60 days after the last dose of AU409 and refrain from donating sperm during this period. WOCBP are eligible to participate if they are not pregnant, not breastfeeding, and agree to follow the contraceptive guidance during the study intervention period and for at least 90 days after the last dose of AU409

  * Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Patients must agree, as part of the informed consent, to undergo liver biopsy (for a subset of patients enrolled at and above dose level 4) and to provide blood for pharmacokinetics analysis
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 8 g/dL (prior transfusion is allowed if completed 2 weeks prior to screening and hemoglobin remains >= 8 g/dL)
* For patients with HCC with splenic sequestration: ANC >= 1000/mm^3
* For patients with HCC with splenic sequestration: Platelets >= 70,000
* Calculated clearance >= 60 mL/min/1.73 m^2. Actual body weight should be used for calculating creatinine clearance (e.g., using the Cockroft-Gault formula). For subjects with a Body Mass Index (BMI) > 30 kg/m^2, lean body weight should be used instead
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (subjects with known Gilbert's hepatic function disease can have bilirubin of up to 2 X ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 X ULN; or AST/ALT =< 5 X ULN if patient has liver tumors
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.8 times upper limit of normal (unless patient is on anticoagulation)

Exclusion Criteria:

* Patients who have had hypersensitivity to pentamidine or any excipients of AU409
* Treatment with other anticancer therapies (including surgery, radiation therapy, chemotherapy, anti-angiogenic therapy, targeted therapy, or radiofrequency ablation therapy, etc.) or investigational therapy within 28 days prior to study entry (except for palliative radiation therapy that should be completed >= 14 days prior to study entry)
* Hepatocellular carcinoma patients with a Child Pugh score >= B7
* Patients with known central nervous system metastases which are untreated or symptomatic; patients with treated brain metastases (completed >= 30 days prior to screening) are allowed provided they are asymptomatic and are off steroids
* Patient with a history of the following within 6 months prior to cycle 1 day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia, cerebrovascular accident, transient ischemic attack, or seizure disorder. Atrial fibrillation is allowed if rate is controlled
* Patients who have corrected QT (QTc) interval to > 470 msec (Fredericia's equation) on 2 out of 3 electrocardiogram (ECG)'s (if first ECG has QTc < 470, no need to repeat, if first ECG has QTc > 470 repeat twice for a total of 3 ECG's)
* Patients who are on therapeutic anticoagulation with warfarin; however, patients on therapeutic doses of with low molecular weight heparins or Factor Xa inhibitors are eligible
* Patient with history of gastrointestinal surgery or malabsorptive conditions that may change the absorption of drugs and/or cause rapid transit (such as total gastrectomy, small bowel resection, etc.)
* Patients who have known active hepatitis B. Patients with chronic hepatitis B who are on anti-viral therapy and have a hepatitis B viral load of =< 500 IU/mL are allowed on the study. Patients with chronic Hepatitis C are allowed
* Patients who have active infection requiring treatment (except hepatitis B and C as noted above) including known human immunodeficiency virus (HIV) infection
* Patients who have concurrent conditions resulting in immune compromise, including chronic treatment with corticosteroids or other immunosuppressive agents
* Patients who have any other condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
* Patients who are on medications that are considered to be strong inducers or inhibitors of the cytochrome P450 isoenzymes should have such medications discontinued or replaced. Such medications should be avoided for one week prior to first dose of treatment and during the trial participation. If these medications are absolutely necessary for the patient and cannot be replaced, enrollment may still be considered on a case by case basis if it is in the patient's best interest and after discussion with the principal investigator (PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2027-03-29 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 28 days
  MTD is defined as the highest dose tested at which none or no more than one patient experienced DLT attributable to the study drug(s), when 6 patients were treated at that dose and are evaluable for toxicity. The MTD is one dose level below the lowest dose tested in which 2 or more patients experienced DLT attributable to the study drug(s.)
Recommended phase II dose | Up to 28 days
  The RP2D for evaluation in Phase 2 will be selected based on overall safety and tolerability, PK, preliminary efficacy, and estimates of efficacious liver exposures extrapolated from nonclinical data and Phase 1 of the study. The RP2D may or may not be the same as the MTD identified in Phase 1. For example, if the MTD was not reached with a plateau of exposures despite increasing drug dose, or if exposure at the MTD was much higher than the level expected to be required for efficacy, or if subsequent cycles of treatment provided additional insight on the safety profile, then the RP2D might be different, though not higher dose than the MTD.
  Additionally, if an MTD is not identified in the dose range expected, a dose that met the tolerability and PK criteria could be selected as the RP2D.
Incidence of adverse events | Up to 30 days after removal from treatment or until death, whichever occurs first
  Will be assessed per Common Terminology Criteria for Adverse Events version 5.0 criteria.

SECONDARY OUTCOMES:
Objective radiologic response | Up 3 years
  Will assess preliminary assessment of anti-tumor activity of AU409 via objective radiologic response using Response Evaluation Criteria in Solid Tumors 1.1 criteria.
Pharmacokinetics evaluation - Peak plasma concentration (Cmax) | Day 1 of cycles 1 and 2. Days 8, 15, and 21 of cycle 1. (cycle = 28 days)
  Pharmacokinetics profile will be evaluated following a comprehensive PK parameter
Pharmacokinetics evaluation - Peak time (Tmax) | Day 1 of cycles 1 and 2. Days 8, 15, and 21 of cycle 1. (Cycle = 28 days)
  Pharmacokinetics profile will be evaluated following comprehensive PK parameter

CONTACTS AND LOCATIONS:
Overall Officials: Anthony B El-Khoueiry, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California